CLINICAL TRIAL: NCT06565559
Title: EMUs: Enhanced Monitoring Using Sensors After Surgery
Acronym: EMUs
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: University of Birmingham (Other); University for Development Studies, Tamale, Ghana (Other); Hospital San Juan de Dios Guatemala (Other Government); Christian Medical College and Hospital, Ludhiana, India (Other); Hospital Español de Veracruz, Veracruz, Mexico (Unknown); University of Rwanda (Other); University of Lagos, Nigeria (Other); School of health sciences, University of Abomey Calavi, Benin (Unknown)
Responsible Party: Sponsor
Other Study IDs: EMUs; 13344828 (Other Grant/Funding Number: Wellcome Leap)
Record Dates: First submitted 2024-07-15; First posted 2024-08-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Surgery; Inpatients
Keywords: Surgery; Wearable Devices; Global Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Study Cohort: All surgical patients that fit the study eligibility criteria.
  Interventions: Device: Wearable Wireless Sensor

INTERVENTIONS:
Device: Wearable Wireless Sensor — Stage III is a shadow mode evaluation of the device with participants wearing sensors pre-, intra-, and post-operatively. Sensor and clinical data will be collected contemporaneously in the clinical environment. No sensor data is made available to clinical teams for decision making, with no change in patient care.

SUMMARY:
Patients can become critically unwell following surgical operations. Delay in recognition of this deterioration can result in patient harm and even death. Wearable wireless sensors that record patients vital signs such as heart rate could help improve recognition of patient deterioration. The goal of this observational study: Enhanced Monitoring Using Sensors After Surgery (EMUs) is to determine if data from wearable physiological monitors can be used for the early detection of postoperative deterioration, while being acceptable to patients and healthcare staff. The study participants and surgical inpatients undergoing open surgery. There are 3 objectives which each represent a stage of the study:

1. To perform usability testing of device with clinicians, nurses, and healthcare workers in non-clinical environment.
2. To determine baseline postoperative monitoring practice across our network and perform device usability testing in clinical environment.
3. To perform a shadow-mode cohort study with collection of time-stamped sensor clinical event data to determine relationships between physiological waveforms and patient deterioration.

This registration focuses on the shadow-mode cohort study.

Participants will wear wireless sensors on their chest and fingers, pre-, intra-, and post-operatively for up to 10 days. The sensors will record their vital signs such as heart rate, and oxygen levels. This will then be analysed, and used to aid the design of early detection algorithms that may be able to predict clinical illness or complications in this patient group. This is an observational study gathering real time data only. No changes in patient care will result, and in Stages 2 and 3 no sensor data will be available to clinical teams. This study will be performed in departments of general surgery in Benin, Ghana, Guatemala, India, Mexico, Nigeria, Rwanda, and the United Kingdom.

DETAILED DESCRIPTION:
Patients who die after surgery frequently have treatable complications which are not identified in a timely manner. This is due to a failure to "recognize", "relay" or "react" to the deterioration of a patient in the postoperative period. This study aims to determine whether data from wearable physiological monitors can be used for the early detection of patient deterioration, while being acceptable to patients and healthcare staff. If found useful, future studies would be conducted to determine the performance and safety of such a device.

This study has three objectives which will be addressed in three stages.

STAGE 1. Usability testing of device with clinicians, nurses, and healthcare workers in non-clinical environment.

STAGE 2. Baseline postoperative monitoring practice assessment and device usability testing in clinical environment.

STAGE 3. Shadow-mode cohort study with collection of time-stamped sensor and clinical event data to determine relationships between physiological waveforms and patient deterioration.

This registration focuses on the shadow-mode cohort study.

This study will be performed in departments of general surgery in Benin, Ghana, Guatemala, India, Mexico, Nigeria, Rwanda, and the UK. In Stages 2 and 3, patients will have undergone major surgery and will be recovering in postoperative wards.

This study can be performed using any suitable wearable device (it is device agnostic), as it seeks to gather generalisable information. In the first instance, the Sibel ANNE® One device will be used. ANNE® One is a wireless ICU-grade dual sensor system that provides real-time physiological monitoring. The system features two skin-mounted, bio-integrated sensors that provide continuous storage of vital sign measurements and physiological waveforms.

This is an observational study gathering real time data only. No changes in patient care will result, and in Stages 2 and 3 no sensor data will be available to clinical teams. True equipoise exists: it is not clear whether these data are useful or how they should be used. Patients will be managed with standard care throughout.

Wearable sensors have potential application in improving postoperative monitoring and consequently, the reduction of avoidable morbidity and mortality. Sensor data may be used to generate prediction algorithms providing a continuous readout of individual patient risk. Such algorithms could enhance healthcare workers' capacity to identify and intervene upon patients with early complications. However, few high-quality studies have yet been performed in this area.

This study has approvals form the following ethical review boards:

Edinburgh Medical School Research Ethics Committee West of Scotland Research Ethics Service (on behalf of NHS Health Research Authority) Health and Care Research Wales (on behalf of NHS Health Research Authority) Ghana Health Service Ethics Review Committee Comite de Investigacion, Hospital General San Juan de Dios, Guatemala, Guatemala Christian Medical College and Hospital, Institutional Ethics Committee, Ludhiana, India El Comite de Etica en Investigacion del Hospital General de Boca del Rio, Veracruz, Mexico Lagos University Teaching Hospital Health Research Ethics Committee, Lagos Nigeria Lagos State University Teaching Hospital Health Research Ethics Committee, Ikeja, Nigeria Obafemi Awolowo University Hospitals Teaching Complex, Ethics and Research Committee, Ife, Nigeria Ethics Committee of University Teaching Hospital of Kigali, Kigali, Rwanda

ELIGIBILITY:
Participant Inclusion Criteria:

* Adults 18 years and older.
* Undergoing an elective or emergency major surgery procedure with a planned skin incision of 5 cm or greater. Any indication for surgery can exist, including benign, malignant, and trauma.
* Willing and able to provide written informed consent.

Participant Exclusion Criteria:

* Those under the age of 18.
* A documented or suspected allergy to adhesive dressings.
* Obstetric patients
* Unwilling or unable to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are all patients undergoing a surgical procedure at the NIHR Global Health Research Unit on Global Surgery hubs/spoke hospitals in India, Nigeria, Ghana, Guatemala, Mexico, Rwanda, Benin and the United Kingdom that fit the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 1332 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular data from wearable device | 0-10 days from device application.
  Data includes core vital sign measures to assess the patient's cardiovascular function (e.g. heart rate in beats per minute), advanced indices (e.g., pulse arrival time, Heart Rate (HR) /Respiratory Rate (RR) quotient) and raw waveform data.
Respiratory data from wearable device | 0-10 days from device application.
  Data includes core vital sign measures to assess the patient's respiratory function (e.g. oxygen saturation as a percentage), advanced indices (e.g, Heart Rate (HR) /Respiratory Rate (RR) quotient) and raw waveform data.
Body temperature data from wearable device | 0-10 days from device application.
  Data includes core vital sign measures (e.g. temperature measurement in degrees centigrade), advanced indices, and raw waveform data.

SECONDARY OUTCOMES:
Standard-of-care cardiovascular vital sign observation data | 0-10 days from day of device application.
  Standard-of-care vital sign observation data to assess cardiovascular function e.g. heart rate in beats per minute, blood pressure in mmHg at a frequency normally collected. These will be assessed as part of the National Early Warning Score 2 system (NEWS2) which a validated early warning score for detecting patient deterioration or equivalent in participating centers.
Standard-of-care respiratory vital sign observation data | 0-10 days from day of device application.
  Standard-of-care vital sign observation data to assess respiratory function e.g. respiratory rate in breaths per minute, oxygen saturations in percentage, at a frequency normally collected. These will be assessed as part of the National Early Warning Score 2 system (NEWS2) which a validated early warning score for detecting patient deterioration, or equivalent in participating centers.
Standard-of-care temperature vital sign observation data | 0-10 days from day of device application.
  Standard-of-care vital sign observation data to assess temperature e.g. in degrees centigrade or Fahrenheit, at a frequency normally collected. These will be assessed as part of the National Early Warning Score 2 system (NEWS2) which a validated early warning score for detecting patient deterioration or equivalent in participating centers.
Standard-of-care neurological observation data | 0-10 days from day of device application.
  Standard-of-care vital sign observation data to assess neurological function e.g. Alert Verbal Pain Unresponsive (AVPU) at a frequency normally collected. These will be assessed as part of the National Early Warning Score 2 system (NEWS2) which a validated early warning score for detecting patient deterioration or equivalent in participating centres.
Incidence of clinical complications during the study period | 0-10 days from the day of device application and then 30 day follow up will be performed.
  Incidence of clinical diagnosis data such as bleeding, major adverse cardiac event, sepsis will be derived from patient records and recorded and any uncertainty reviewed post hoc by an expert adjudication panel. Clinical complication data will also be gathered at 30 days.
Incidence of clinical investigations during the study period | 0-10 days from the day of device application.
  The incidence of clinical investigations and descriptive details about the investigations will be derived from the patient records such as chest xray, CT abdomen, and wound swab.
Incidence of clinical interventions during the study period | 0-10 days from the day of device application.
  The incidence of clinical interventions performed and descriptive details, during the period of the device being worn will be recorded, e.g. commencement of antibiotics, unplanned admission to critical care, unplanned reoperation.
Incidence and results of blood tests to assess patient physiological status during the study period | 0-10 days from the day of device application.
  The incidence of blood tests will be recorded and the associated results from during the 10 day study period. Bloods tests recorded will include full blood count, urea and electrolytes, inflammatory markers, liver function tests and coagulation profile as well as blood gas results. They will be recorded using whichever the standard units are at participating centres.

CONTACTS AND LOCATIONS:
Overall Officials: Ewen Harrison, Principal Investigator — University of Edinburgh
Locations (17):
- Benin (4):
  - Hopital de Zone Atlantique Ouidah, Ouidah, Atlantique Department
  - Centre Hospitalier Universitaire Departemental Borgou-Alibori, Parakou, Borgou Department
  - Centre Hospitalier Universitaire Mere Enfant Lagune, Cotonou, Littoral Department
  - Centre Hospitalier Universitaire et Departemental Oueme Plateau, Porto-Novo, Oeume
- Ghana (3):
  - Berekum Holy Family Hospital, Berekum, Berekum East
  - Techiman Holy Family Hospital, Techiman, Bono East
  - Tamale Teaching Hospital, Tamale
- Hospital General San Juan de Dios, Guatemala City, Guatemala
- India (3):
  - Lady Willingdon Hospital, Manali, Himachal Pradesh
  - Padhar Hospital, Pādhar, Madhya Pradesh
  - Christian Medical College and Hospital, Ludhiana, Punjab
- Hospital Español de Veracruz, Veracruz, Mexico
- Nigeria (3):
  - Obafemi Awolowo University Teaching Hospital Complex, Ife
  - Lagos State University Teaching Hospital, Ikeja
  - Lagos University Teaching Hospital, Lagos
- University Teaching Hospital of Rwanda, Kigali, Rwanda
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

REFERENCES:
- [Background] Burke JR, Downey C, Almoudaris AM. Failure to Rescue Deteriorating Patients: A Systematic Review of Root Causes and Improvement Strategies. J Patient Saf. 2022 Jan 1;18(1):e140-e155. doi: 10.1097/PTS.0000000000000720. PMID 32453105
- [Background] Ghaferi AA, Birkmeyer JD, Dimick JB. Variation in hospital mortality associated with inpatient surgery. N Engl J Med. 2009 Oct 1;361(14):1368-75. doi: 10.1056/NEJMsa0903048. PMID 19797283
- [Derived] Jiwa A, Cameron MM, Ademuyiwa AO, Adisa A, Aguilera Arevalo ML, Bahrami Hessari M, Bhangu A, Brennan PM, Clark N, Cresswell K, Czerwinska I, D'Adderio L, Gunn E, Haque PD, Ikegwuonu T, Lawani I, Morton D, Nganwa A, Ntirenganya F, Pius R, Ramos de la Medina A, Samuel S, Shaw CA, Tabiri S, Townsend RC, Varghese C, Ghosh D, Harrison EM; NIHR Global Health Research Unit on Global Surgery. Continuous physiological monitoring for the detection of postoperative deterioration: a protocol for a multistage, multicentre, international, prospective cohort study. BMJ Open. 2025 Oct 6;15(10):e104463. doi: 10.1136/bmjopen-2025-104463. PMID 41057181